CLINICAL TRIAL: NCT06722768
Title: Identifying Gait Changes From a Cerebrospinal Fluid Tap Test Using a Smart Insole in Idiopathic Normal Pressure Hydrocephalus
Brief Title: Identifying Gait Changes From a CSF Tap Test Using a Smart Insole in iNPH
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 9-2024-0130
Record Dates: First submitted 2024-11-27; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: gait analysis; smart insole; Cerebrospinal fluid tap test
MeSH Terms: conditions — Hydrocephalus, Normal Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responder group: Patients with iNPH were divided into responder group and non-responder group after CSF tap test.
  The responder group consists of patients who underwent the tap test and exhibited improvements in gait and balance, including increased gait speed as measured by the 10-Meter Walk Test (10MWT), reduced time on the Timed Up and Go Test (TUGT), and resolution of shuffling, magnetic, and wide-based gait patterns. Classification were done by a multidisciplinary team including physiatrist, neurologist, and neurosurgeon.
  Surgical treatment was carefully considered for the responder group. Patients who declined surgery or were considered at high risk for surgical complications due to advanced age or comorbidities were excluded. Patients who were able to get an operation primarily underwent shunt surgery.
  Additional gait and balance analyses were performed on patients who underwent surgery within 24 hours after their last operation.
- Non-Responder group: Patients with iNPH were divided into responder group and non-responder group after CSF tap test.
  The non-responder group consists of patients who underwent the tap test but did not exhibit improvements in gait or balance. Classification were done by a multidisciplinary team including physiatrist, neurologist, and neurosurgeon.
  Surgical treatment was not considered for the responder group.

SUMMARY:
The goal of this clinical trial is to to evaluate various gait parameters by a sensor-embedded smart insole before and after the cerebrospinal fluid (CSF) tap test in idiopathic normal pressure hydrocephalus (iNPH) patients.

The main questions it aims to answer are:

* Does the CSF tap test enhance gait and balance parameters in participants?
* Does the CSF tap test enhance cognitive and urinary symptoms in participants?

Researchers will compare pre- and post-CSF tap test gait and balance parameters by a sensor-embedded smart insole.

Participants will:

* Participate in physical function assessments including the 10-meter walk test, Timed Up and Go test, and Berg Balance Scale wearing sensor-embedded smart insoles before and after the CSF tap test.
* Complete survey about cognitive and unary symptoms before and after the CSF tap test.

DETAILED DESCRIPTION:
Patients who were diagnosed as probable iNPH and underwent CSF tap test at Yongin Severance Hospital, Korea between June 2021 and October 2024 enrolled to our study. Patients were considered as probable iNPH when both satisfying clinical criteria and radiologic criteria All patients underwent a spinal CSF tap test draining 30mL of CSF. Surgical treatment was considered for patients who positively responded to CSF tap test. All patients gave their informed consent to participation in the study.

Gait and balance were assessed both in pre-24 hr of CSF tap test and post-24 hr of CSF tap test. Additional analyses were performed on patients who underwent surgery.

Timed-up-and go Test (TUGT) and 10-meter walk Test (10MWT) were done to evaluate the gait of patients. TUGT timed how long it took participant to stand up, go 3 meters, turn around, come back 3 meters, and sit down. 10MWT calculated walking speed by dividing 10 meters by the time taken to walk the distance. These two tests were recorded and stored as a video. The Balance was assessed through Berg Balance Score (BBS). BBS evaluated set of 14 balance related tasks and scores out of 56 points.

The spatiotemporal gait parameters and data stream of plantar pressure and acceleration were investigated during 10MWT. The patients wore commercial smart insoles with embedded four pressure sensors and three-axis accelerometers (GDCA-MD®,Gilon, Republic of Korea) during 10MWT. It measures real-time plantar pressure in four areas of the foot(toe, lateral midfoot, medial midfoot, and heel) and three-axis acceleration and displays them on a tablet with automatically calculated spatiotemporal gait parameters(step count, cadence, stride length, stride time, swing ratio).

Cognitive and Urinary symptoms were assessed at the baseline. Mini-Mental State Examination (MMSE) was done to measure neuropsychological status. Urinary symptom was graded based on the Overactive Bladder Symptom Score(OABSS) and International Prostate Symptom Score(IPSS).

ELIGIBILITY:
Inclusion Criteria:

* individuals who have more than 1 symptom in the clinical triad including gradually developed gait disturbances mainly showing shuffling, magnetic, wide based gait
* individuals who assessed a standardized cranial MRI scan and those with an Evans ratio greater than 0.30 were included in the study (Microvascular lesions in the white matter were accepted only if they were mild.)
* individuals who voluntarily agree to participate in the study and sign a consent form

Exclusion Criteria:

* individuals with history of hemorrhage
* individuals unable to walk independently on flat ground for 10 meters
* individuals with clinically significant disorders in the cardiovascular, gastrointestinal, respiratory, or endocrine systems
* individuals considered clinically unsuitable for the trial by the trial manager or person in charge based on significant medical findings

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Single general hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Timed up and go test (TUG) | This session will be performed at baseline and at end-point. A baseline assessment will be conducted within 24 hours before the CSF tap test, and an end-point assessment will be conducted within 24 hours after the CSF tap test.
  Researchers ask patients to rise from a seated position, walk a distance of 3 m, turn around, return to the chair, and sit back. The average time of three trials was recorded as a result.
10 meter walk test (10MWT) | This session will be performed at baseline and at end-point. A baseline assessment will be conducted within 24 hours before the CSF tap test, and an end-point assessment will be conducted within 24 hours after the CSF tap test.
  Patients are instructed to walk 14 m, including 2 m at both ends for acceleration and deceleration, at their comfortable speed. Gait speed was calculated by dividing the 10m distance by the time taken.
Berg balance scale (BBS) | This session will be performed at baseline and at end-point. A baseline assessment will be conducted within 24 hours before the CSF tap test, and an end-point assessment will be conducted within 24 hours after the CSF tap test.
  Patients are asked to perform 14 tasks regarding the static and dynamic balance of patients. Each task was rated on a five-point scale from 0 to 4, with a total score of 56.
Total steps of walking | This session will be performed at baseline and at end-point. A baseline assessment will be conducted within 24 hours before the CSF tap test, and an end-point assessment will be conducted within 24 hours after the CSF tap test.
  Spatiotemporal parametric data of gait collected while the subject is performing a home-based activity wearing an insole, recording total steps.
Cadence of walking | This session will be performed at baseline and at end-point. A baseline assessment will be conducted within 24 hours before the CSF tap test, and an end-point assessment will be conducted within 24 hours after the CSF tap test.
  Spatiotemporal parametric data of gait collected while the subject is performing a home-based activity wearing an insole, recording steps per minute.
Velocity of walking | This session will be performed at baseline and at end-point. A baseline assessment will be conducted within 24 hours before the CSF tap test, and an end-point assessment will be conducted within 24 hours after the CSF tap test.
  Spatiotemporal parametric data of gait collected while the subject is performing a home-based activity wearing an insole, recording gait speed (km/h).
Stride length of walking | This session will be performed at baseline and at end-point. A baseline assessment will be conducted within 24 hours before the CSF tap test, and an end-point assessment will be conducted within 24 hours after the CSF tap test.
  Spatiotemporal parametric data of gait collected while the subject is performing a home-based activity wearing an insole, recording stride length (m).
Stride time of walking | This session will be performed at baseline and at end-point. A baseline assessment will be conducted within 24 hours before the CSF tap test, and an end-point assessment will be conducted within 24 hours after the CSF tap test.
  Spatiotemporal parametric data of gait collected while the subject is performing a home-based activity wearing an insole, recording stride time (s).
Swing phase rate of walking | This session will be performed at baseline and at end-point. A baseline assessment will be conducted within 24 hours before the CSF tap test, and an end-point assessment will be conducted within 24 hours after the CSF tap test.
  Spatiotemporal parametric data of gait collected while the subject is performing a home-based activity wearing an insole, recording swing phase rate (%).
Mean peak pressure | This session will be performed at baseline and at end-point. A baseline assessment will be conducted within 24 hours before the CSF tap test, and an end-point assessment will be conducted within 24 hours after the CSF tap test.
  The insole raw data stream was analyzed as following process. Pressure sensor measured foot pressure 40 times per second as relative values (0∼1,023). We obtained periodic foot pressure graphs for each foot region. From these graphs, mean peak pressure were determined by splitting the graph for each step, identifying the maximum pressure value in each step, and averaging the peak pressure values. The relative pressure values were subsequently converted into kilopascals using a validated algorithm with the conversion formula.

SECONDARY OUTCOMES:
Korean Mini-Mental State Examination | This session will be performed at baseline and at end-point. A baseline assessment will be conducted within 24 hours before the CSF tap test, and an end-point assessment will be conducted within 24 hours after the CSF tap test.
  A test that assesses the degree of overall cognitive impairment, taking into account a person's level of education, and the test assesses time and place perception, attention and calculation, memory, language, and spatial and temporal organization. The examiner asks questions corresponding to the items on the test sheet below and record a score for the answers.
Overactive Bladder Symptom Score | This session will be performed at baseline and at end-point. A baseline assessment will be conducted within 24 hours before the CSF tap test, and an end-point assessment will be conducted within 24 hours after the CSF tap test.
  Questionnaire designed to assess the severity of overactive bladder symptoms and their impact on patients' quality of life.
International Prostate Symptom Score | This session will be performed at baseline and at end-point. A baseline assessment will be conducted within 24 hours before the CSF tap test, and an end-point assessment will be conducted within 24 hours after the CSF tap test.
  Questionnaire designed to evaluate the severity of lower urinary tract symptoms commonly associated with benign prostatic hyperplasia. It also assesses the impact of these symptoms on the patient's quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Yongin Severance Hospital, Yongin-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shprecher D, Schwalb J, Kurlan R. Normal pressure hydrocephalus: diagnosis and treatment. Curr Neurol Neurosci Rep. 2008 Sep;8(5):371-6. doi: 10.1007/s11910-008-0058-2. PMID 18713572
- [Background] Kiefer M, Unterberg A. The differential diagnosis and treatment of normal-pressure hydrocephalus. Dtsch Arztebl Int. 2012 Jan;109(1-2):15-25; quiz 26. doi: 10.3238/arztebl.2012.0015. Epub 2012 Jan 9. PMID 22282714
- [Background] Halperin JJ, Kurlan R, Schwalb JM, Cusimano MD, Gronseth G, Gloss D. Practice guideline: Idiopathic normal pressure hydrocephalus: Response to shunting and predictors of response: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology. Neurology. 2015 Dec 8;85(23):2063-71. doi: 10.1212/WNL.0000000000002193. PMID 26644048
- [Background] Dias SF, Graf C, Jehli E, Oertel MF, Mahler J, Schmid Daners M, Stieglitz LH. Gait pattern analysis in the home environment as a key factor for the reliable assessment of shunt responsiveness in patients with idiopathic normal pressure hydrocephalus. Front Neurol. 2023 Apr 4;14:1126298. doi: 10.3389/fneur.2023.1126298. eCollection 2023. PMID 37082443
- [Background] Stolze H, Kuhtz-Buschbeck JP, Drucke H, Johnk K, Diercks C, Palmie S, Mehdorn HM, Illert M, Deuschl G. Gait analysis in idiopathic normal pressure hydrocephalus--which parameters respond to the CSF tap test? Clin Neurophysiol. 2000 Sep;111(9):1678-86. doi: 10.1016/s1388-2457(00)00362-x. PMID 10964082
- [Background] Jang CW, Park K, Paek MC, Jee S, Park JH. Validation of the Short Physical Performance Battery via Plantar Pressure Analysis Using Commercial Smart Insoles. Sensors (Basel). 2023 Dec 11;23(24):9757. doi: 10.3390/s23249757. PMID 38139603